CLINICAL TRIAL: NCT00415337
Title: Endobronchial Ultrasound Guided Transbronchial Lung Biopsy With or Without Guide Sheath in Lung Tumors and the Analysis of Echoic Patterns of Lung Tumors and Mediastinal Lymph Nodes, and the Association Between Diagnostic Yield of Transbronchial Lung Biopsy and EBUS Echoic Features.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHIH-HSI KUO, MD, Chang Gung Memorial Hospital
Other Study IDs: ebus101101
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Lung Neoplasms
Keywords: lung; neoplasm; bronchoscopy; ultrasonography; histology
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort

INTERVENTIONS:
Procedure: endobronchial ultrasound — EBUS

SUMMARY:
1. Endobronchial ultrasonography (EBUS) is useful in localizing peripheral lung lesions. The EBUS, further combined with the guide sheath (GS) technique, has been reported to increase the yield of transbronchial biopsy. However, there are no reports comparing the GS technique and the traditional EBUS technique in diagnosing the peripheral lung tumor.
2. Previous reports have revealed that several characteristic echoic patterns correlate well with the histopathological findings of benign and malignant lesions. Therefore, EBUS may also be useful in the differential diagnosis of malignant lesions of the lung.

ELIGIBILITY:
Inclusion Criteria:

* Patient with radiologically confirmed peripheral lung mass

Exclusion Criteria:

* Patient clinically not indicated for bronchoscopy exam within the abovementioned cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with radiologically confirmed peripheral lung mass
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Han-Pin Kuo, Chair, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taipei, Taiwan